CLINICAL TRIAL: NCT07229768
Title: A Single-Center, Single-Arm, Open-Label Clinical Study of 177Lu-CTR-FAPI Injection in the Treatment of Patients With Advanced, Metastatic Solid Tumors
Brief Title: Clinical Study of 177Lu-CTR-FAPI In the Treatment of Patients With Advanced, Metastatic Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yan Xing (Other)
Responsible Party: Sponsor-Investigator, Yan Xing, Medical Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025-139
Record Dates: First submitted 2025-09-29; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-CTR-FAPI Treatment Arm (Experimental)
  Interventions: Drug: 177Lu-CTR-FAPI

INTERVENTIONS:
Drug: 177Lu-CTR-FAPI — The medication is administered intravenously, with a single dose of 200 mCi (7.4 GBq) ±10%, administered once every 6 ± 2 weeks. The planned course consists of 4 doses, or until the radiation safety threshold for major organs is reached based on radiation dosimetry assessment.

SUMMARY:
This is a single-center, single-arm, open-label clinical study of 177Lu-CTR-FAPI injection in the treatment of patients with advanced, metastatic solid tumors i.e. pancreatic cancer, to assess safety, radio-dosimetry, and efficacy per RESIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients with unresectable, advanced, or metastatic solid tumors who have been histologically or cytologically confirmed, have failed standard treatment, lack standard treatment options, or refuse standard treatment. Preferred tumor types include pancreatic cancer, breast cancer, and soft tissue sarcoma, and must meet any of the following tumor-specific criteria:

  1. Patients with advanced or metastatic TNBC who have progressed after or are intolerant to at least 2 lines of systemic therapy;
  2. Patients with HER2-positive advanced or metastatic breast cancer who have progressed after or are intolerant to at least 2 lines of HER2-targeted therapy;
  3. Patients with HR/HER2-negative advanced or metastatic breast cancer who have progressed after or are intolerant to at least 2 lines of systemic therapy;
  4. Patients with advanced or metastatic high-grade soft tissue sarcoma (excluding chordoma) who have progressed after or are intolerant to at least 1 line of systemic therapy;
  5. Patients with advanced or metastatic pancreatic cancer who have progressed after or are intolerant to at least 1 line of systemic therapy.
* 2: Age >= 18 years, regardless of sex;
* 3: Able to understand and sign informed consent and willing and able to comply with study and follow-up procedures;
* 4: ECOG performance status score of 0 or 1;
* 5: FAP expression in tumor lesions confirmed positive by FAPI PET/CT;
* 6: Agree to provide archived or fresh tumor tissue for immunohistochemical evaluation (if available);
* 7: At least 1 measurable lesion according to RECIST 1.1 criteria;
* 8: Previous anti-tumor toxicities recovered to grade 0-1;
* 9: Organ function meets requirements before first administration;

  1. Hematology: Absolute neutrophil count (ANC) >= 1.5×10^9/L; Hemoglobin (Hb) >= 80 g/L; Platelet count (PLT) >= 75×10^9/L;
  2. Liver function: Total bilirubin (TB) <= 1.5×ULN; AST and ALT <= 3×ULN, and if there is hepatic tumor metastasis, ALT and AST <= 5×ULN;
  3. Renal function: Creatinine clearance >= 50 mL/min (Cockcroft-Gault formula); ECG: QTcF <= 470 ms;
* 10: Fertile subjects voluntarily use effective contraception during treatment and for 4 months (male) or 7 months (female) after the last dose of study drug.

Exclusion Criteria:

* 1: Subjects with brain metastases, meningiomas, or other central nervous system lesions at screening
* 2: Severe allergy to contrast agents or claustrophobia
* 3: Expected survival period < 6 months
* 4: Receipt of blood transfusion within 2 weeks before the first dose to meet the eligibility criteria
* 5: Administration of systemic antitumor therapies (including targeted therapy, immunotherapy, traditional Chinese medicine antitumor treatment, chemotherapy, etc.) within 4 weeks prior to the first dose
* 6: Participation in other clinical trials involving investigational drugs or devices within 4 weeks before the first dose
* 7: Major surgery within 4 weeks before the first dose or planned major surgery during the study period
* 8: Active bacterial, fungal, viral, or other infections requiring intravenous medication within 4 weeks before the first dose
* 9: Previous systemic radionuclide therapy (excluding I-131 treatment for thyroid cancer) or external beam radiotherapy (EBRT) within 4 weeks prior to the first dose
* 10: History of other malignancies within 5 years before the first dose
* 11: Severe cardiovascular or cerebrovascular diseases, or poorly controlled diabetes
* 12: Presence of pleural effusion or ascites requiring treatment or judged by the investigator as uncontrolled at screening
* 13: Females who are pregnant or breastfeeding
* 14: Subjects considered by the investigator to have poor compliance and inability to cooperate with treatment and follow-up at screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AE | From enrolment to 12 months after the first dose
  Adeverse Events

SECONDARY OUTCOMES:
Radiation Dosimetry | one week after first dose
ORR | From first dose to 12 months afer
  Objective Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No